CLINICAL TRIAL: NCT04560049
Title: Comparison of Phenol and Silver Nitrate Application in the Sacrococcygeal Pilonidal Sinus: A Prospective Randomized Controlled Study
Brief Title: Phenol and Silver Nitrate Application in Pilonidal Sinus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hanife Seyda Ulgur, Assistant Doctor, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/206
Record Dates: First submitted 2020-09-09; First posted 2020-09-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pilonidal Sinus of Natal Cleft; Pilonidal Sinus Without Abscess
Keywords: Pilonidal Sinus; Phenol; Silver Nitrate
MeSH Terms: conditions — Pilonidal Sinus | interventions — Silver Nitrate; Phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenolisation (Experimental): Surgical pit excision and phenolisation of sinus tract
  Interventions: Drug: Phenol
- Silver Nitrate Irrigation (Active Comparator): Surgical pit excision and silver nitrate irrigation of sinus tract
  Interventions: Drug: Silver Nitrate

INTERVENTIONS:
Drug: Silver Nitrate — application of silver nitrate to sinus tract
  Arms: Silver Nitrate Irrigation
Drug: Phenol — phenolisation of sinus tract
  Arms: Phenolisation

SUMMARY:
Pilonidal sinus is a disease that affects the young population. Wound healing is a problem after surgical interventions Especially wound healing brings minimally invasive interventions to the fore. In this study we will administer two types of irritating agent for pilonidal sinus disesase. One of them is phenol and second one is silver nitrate solution. And not routinely used for pilonidal sinus disease. The data about availeble in pubmed and google scholar is limited focused on silver nitrate The goal of the study is to compare the silver nitrate and phenol application

DETAILED DESCRIPTION:
Sacrococcygeal pilonidal sinus disease is a chronic subcutaneous tissue inflammation that most commonly affects the male sex between the ages of 20 and 30, characterized by burning, itching and discharge in the internal gluteal cleft. It affects the young working population, short return to work after treatment and early return to daily normal activity is socioeconomically important. Although approximately 15 different surgical techniques have been described in the literature in the treatment of pilonidal sinus, a gold standard approach has not been determined. Since it is seen in the young working population, it is important that the ideal treatment has an easy-to-apply, low cost and fast recovery process. The effectiveness of phenol administration as a minimally invasive procedure has been demonstrated with acceptable complication and success rates in prospective and retrospective studies.

Silver nitrate is a caustic and sclerosing substance that impairs tract integrity, such as phenol. It supports the closure of the sinus tract by cauterizing the granulation and epithelialized tissue throughout the sinus. It also has antimicrobial properties to reduce microbial load throughout the tract. Although the effective use and successful results of silver nitrate in the treatment of perianal fistula have been shown, a prospective study has not been conducted yet on the use of pilonidal sinus.

The main purpose of the study is to compare return to normal daily activity between the two groups. This period will be measured in days from the intervention. Participants will not be offered any restrictions after the intervention, and the period of returning to normal daily activities such as starting work at work or doing the housework will be determined by filling out a two-week daily questionnaire. Secondary goals; quality of life, complaints related to pilonidal sinus (itching, burning, discharge), wound infection, closure of pilonidal sinus mouth, recurrence rate and VAS (visual analog scale) scoring.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients who applied to general surgery outpatient clinic for chronic sacrococcygeal pilonidal sinus
* Patients with written informed voluntary consent forms.

Exclusion Criteria:

* BMI > 35 kg/m²
* Recurrent cases
* Active abscess formation
* Patients with hydradenitis suppurativa and skin lesions in the perianal region
* Patients with accompanying anal fistula, anal conduloma and perianal involvement of Crohn's disease
* Immunosuppressive patients (HIV +, organ transplantation, patients receiving immunosuppressive therapy)
* Complicated cases (have more than 3 orifice)
* Patients with known allergic sensitivity to one of the silver nitrate, phenol, nitrofurazone and prilocaine substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Healing of the pilonidal sinus disease | 8 week
  Closure of pit without pus and soiling on physical examination

SECONDARY OUTCOMES:
Post-procedure Quality of life assessment | 3rd and 8th week after the procedure
  The quality of life of the patients will be determined by SF-36 test.
Wound infection | 3rd and 8th week after the procedure
  Wound infection is simply classifed as present or not present. It is considered as present when there was a an odd smelling purulent discharge from the wound.
Visual analog scale as pain assessment | 3rd and 8th week after the procedure
  Pain of the patients will be determined by VAS (visual analog scale). Patients are simply asked to score their pain from 1 to 10, which is typically called visual analog scale in the literature, with higher scores representing more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Ş Ülgür, Principal Investigator — University of Health Sciences Umraniye Education and Research Hospital
Locations (1):
- University of Health Sciences Umraniye Education and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Result] Pronk AA, Smakman N, Furnee EJB. Short-term outcomes of radical excision vs. phenolisation of the sinus tract in primary sacrococcygeal pilonidal sinus disease: a randomized-controlled trial. Tech Coloproctol. 2019 Jul;23(7):665-673. doi: 10.1007/s10151-019-02030-w. Epub 2019 Jul 5. PMID 31278458
- [Result] Attaallah W, Tuney D, Gulluoglu BM, Ugurlu MU, Gunal O, Yegen C. Should we consider topical silver nitrate irrigation as a definitive nonsurgical treatment for perianal fistula? Dis Colon Rectum. 2014 Jul;57(7):882-7. doi: 10.1097/DCR.0000000000000143. PMID 24901690
- [Result] Kayaalp C, Aydin C. Review of phenol treatment in sacrococcygeal pilonidal disease. Tech Coloproctol. 2009 Sep;13(3):189-93. doi: 10.1007/s10151-009-0519-x. Epub 2009 Aug 5. PMID 19655223
- [Result] Emiroglu M, Karaali C, Esin H, Akpinar G, Aydin C. Treatment of pilonidal disease by phenol application. Turk J Surg. 2017 Mar 1;33(1):5-9. doi: 10.5152/UCD.2016.3532. eCollection 2017. PMID 28589180